CLINICAL TRIAL: NCT02798926
Title: Polyethylene Bag: a Way of Preventing Hypothermia During Central Venous Catheter Placement in Preterm Neonates?
Acronym: PSac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: AOL09-DR-GHYSELEN
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Preterm Neonates
Keywords: hypothermia; central venous catheter placement; Polyethylene bag
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- with the use of a polyethylene bag
  Interventions: Device: polyethylene bag
- without the use of a polyethylene bag

INTERVENTIONS:
Device: polyethylene bag — The infant will be wrapped in a polyethylene bag 15 min before starting central venous catheter placement
  Groups: with the use of a polyethylene bag

SUMMARY:
Particular attention is paid to thermal management of preterm neonates in neonatal intensive care units because of the major risk of morbidity associated with hypothermia. Percutaneous central venous catheter placement is essential to ensure adequate caloric intake and intravenous administration of treatments, but this procedure can cause major body temperature variations, responsible for complications in these neonates, as convection incubator function is impaired during opening of the incubator, which can be prolonged (30 minutes to 2 hours) depending on the technical difficulties encountered during catheter placement.

In parallel, the use of a polyethylene bag or sheet in the delivery room and for neonatal transport is now clearly defined and ensures stability or even a considerable temperature gain during transfer immediately after birth. In the light of several clinical cases, the use of a polyethylene bag during central venous catheter placement appears to be effective to prevent body temperature loss in preterm neonates. No data are currently available concerning the value of this method of prevention of hypothermia during this type of procedure.

Preliminary studies conducted by our team on a dummy suggest that a polyethylene bag or sheet could be useful during this procedure by significantly reducing heat loss caused by convection and evaporation. However, compensation phenomena such as generalized vasoconstriction to cold in preterm infants are very poorly described, but can induce a functional conflict between mechanisms ensuring maintenance of homeostasis and those involved in maintenance of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* premature Newborn child = 32 weeks of gestational age
* 7 days of life
* Normothermic (core temperature between 36.5 and 37.5 ° C)
* Stable on a hemodynamically manner
* Need the installation of a central catheter KTEC

Exclusion Criteria:

* Parental Refusal
* hypothermia (temperature < 36.5 ° C)
* Hyperthermia (temperature > 37.5 ° C)
* heart disease and malformation syndromes life-threatening
* Hemodynamic instability ( catecholamine vasoconstrictor and vasodilator )
* Breakdown by oscillation

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm neonates less than 32 weeks of gestational age (WGA)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Temperature | 1 hour
  difference between the prehepatic temperature at the beginning of catheter placement and the lowest temperature observed during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GHYSELEN, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France